CLINICAL TRIAL: NCT00352963
Title: Study to Assess Immunogenicity and Reactogenicity of Three Doses of GSK Bio's Combined Hib-MenC Vaccine Co-admind With GSK Bio's DTPa-HBV-IPV Vaccine and of Two Doses of Baxters Meningococcal C Conjugate Vaccine Co-admind With GSK Bio's DTPa-HBV-IPV/Hib Vaccine
Brief Title: Immunogenicity & Safety Study of Combined/Separate Vaccine(s) Against Common Diseases in Infants (2,4,6 Months of Age).
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 217744/097
Record Dates: First submitted 2006-07-14; First posted 2006-07-17 (Estimated); Last update posted 2020-01-06 (Actual); Status verified 2020-01

CONDITIONS: Poliomyelitis; Tetanus; Acellular Pertussis; Hepatitis B; Diphtheria
Keywords: Open, phase 3, Infanrix hexa™, Hib-MenC, co-administered
MeSH Terms: conditions — Poliomyelitis; Tetanus; Hepatitis B; Diphtheria

INTERVENTIONS:
Biological: Study vaccines: IH+Hib-MenC/NVC; Control: IH+Meningitec

SUMMARY:
This study will evaluate the immunogenicity of the co-administration of different combinations of DTPa, IPV, hepatitis B, Hib and Men C vaccines during the first year of life.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female infant between, & including, 0 & 7 days of age at the time of the inclusion. Born after a normal gestation period (between 36 & 42 weeks).
* Written informed consent obtained from the parent/guardian of the subject.

Exclusion Criteria:

* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine(s) or planned use during the study period.
* Administration of immunosuppressants or other immune-modifying drugs from birth.
* Administration of immunoglobulins and/or any blood products since birth or planned administration during the study period.
* Administration / planned administration of a vaccine not foreseen by the study protocol during the period starting from birth and ending 30 days after the last dose except BCG vaccination if given before the 30-day period preceding the administration of the 1st dose of Infanrix penta™ or Infanrix hexa™ in combination with a meningococcal C vaccine.
* Evidence of previous or intercurrent diphtheria, tetanus, pertussis, polio, hepatitis B, meningococcal C and Hib disease.
* Evidence of previous diphtheria, tetanus, pertussis, polio, hepatitis B, meningococcal C and Hib vaccination.

Max Age: 7 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 480 (Actual)
Dates: Start 2003-09-30 (Actual); Study Completion 2004-07-16 (Actual)

PRIMARY OUTCOMES:
At M7: Antibodies to PRP, MenC HBsAg

SECONDARY OUTCOMES:
At M7: Abs. to all vaccine antigens
At M6: Abs. to PRP & MenC
Solicited (D0-3); unsol. events (D0-30); SAEs (full study)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (17):
- Spain (17):
  - GSK Investigational Site, Alcorcón
  - GSK Investigational Site, Almeira
  - GSK Investigational Site, Badalona
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Bilbao
  - GSK Investigational Site, Burgos
  - GSK Investigational Site, Córdoba
  - GSK Investigational Site, Getafe
  - GSK Investigational Site, Leganés
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Marid
  - GSK Investigational Site, Málaga
  - GSK Investigational Site, Móstoles/Madrid
  - GSK Investigational Site, Palma de Mallorca
  - GSK Investigational Site, Seville
  - GSK Investigational Site, Valladolid
  - GSK Investigational Site, Vélez-Málaga

IPD SHARING:
Plan to Share IPD: Yes
IPD is available via the Clinical Study Data Request site (click on the link provided below)
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com/Posting.aspx?ID=337

REFERENCES:
- [Background] Tejedor JC, Moro M, Ruiz-Contreras J, Castro J, Gomez-Campdera JA, Navarro ML, Merino JM, Martin-Ancel A, Roca J, Garcia-del-Rio M, Jurado A, Diez-Delgado FJ, Omenaca F, Garcia-Sicilia J, Boceta R, Garcia-Corbeira P, Jacquet JM, Collard A, Schuerman L; Spanish DTaP-HBV-IPV-097 Study Group. Immunogenicity and reactogenicity of primary immunization with a hexavalent diphtheria-tetanus-acellular pertussis-hepatitis B-inactivated polio-Haemophilus influenzae type B vaccine coadministered with two doses of a meningococcal C-tetanus toxoid conjugate vaccine. Pediatr Infect Dis J. 2006 Aug;25(8):713-20. doi: 10.1097/01.inf.0000227725.61495.c4. PMID 16874171
- [Background] Tejedor JC, Moro M, Ruiz-Contreras J, Castro J, Gomez-Campdera JA, Navarro ML, Merino JM, Martin-Ancel A, Roca J, Garcia-Del-Ri M, Jurado A, Diez-Delgado FJ, Omenaca F, Garcia-Sicilia J, Boceta R, Garcia-Corbeira P, Collard A, Boutriau D, Schuerman L, Jacquet JM; Spanish DTPa-HBV-IPV-097 Study Group. Immunogenicity and reactogenicity of primary immunization with a novel combined Haemophilus influenzae Type b and Neisseria meningitidis Serogroup C-tetanus toxoid conjugate vaccine coadministered with a Diphtheria-tetanus-acellular Pertussis-hepatitis B-inactivated poliovirus vaccine at 2, 4 and 6 months. Pediatr Infect Dis J. 2007 Jan;26(1):1-7. doi: 10.1097/01.inf.0000247070.60063.09. PMID 17195697
- [Background] Jeanne Jaquet et al. Co-administration of DTPa-HBV-IPV/Hib with two doses of a MenC-TT conjugate vaccine in primary vaccination - 23rd Annual Meeting ESPID, Valencia, Spain, 18-20 May 2005.
- [Background] Tejedor et al. Immunogenicity and reactogenicity of a novel combined Haemophilus influenzae type b and Neisseria meningitidis serogroup C-tetanus toxoid conjugate (Hib-MenC-TT) Vaccine co-administered with a pentavalent DTPa-HBV-IPV vaccine at 2, 4 and 6 months - 24th Annual Meeting ESPID, Basel, Switzerland, 03-05 May 2006.
- [Background] Tozzi AE, Azzari C, Bartolozzi G, Esposito S, Fara GM, Giudice ML. Can hexavalent vaccines be simultaneously administered with pneumococcal or meningococcal conjugate vaccines? Hum Vaccin. 2007 Nov-Dec;3(6):252-9. doi: 10.4161/hv.4626. Epub 2007 Jun 23. PMID 17881905
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Clinical Study Report: 217744/097 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 217744/097 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 217744/097 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 217744/097 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 217744/097 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 217744/097 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register